CLINICAL TRIAL: NCT06556849
Title: Effectiveness of Defocus Incorporated Multiple Segments in Slowing Myopia Progression as a Function of the Age in Pediatric Patients. Three Years Follow up.
Brief Title: Effectiveness of DIMS Spectacle as a Function of the Age
Status: Completed | Type: Observational
Sponsor: Luca Buzzonetti (Other)
Responsible Party: Sponsor-Investigator, Luca Buzzonetti, Head of Ophthalmology Unit, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Other Study IDs: Myopia1
Record Dates: First submitted 2024-07-19; First posted 2024-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: patients oldest than 10 years that wear DIMS lens: myopic patients oldest than 10 years of age that wore Defocus Incorporated Multiple Segments (DIMS) spectacles
  Interventions: Device: Defocus Incorporated Multiple Segments (DIMS)
- Group B: patients oldest than 10 years that wear (control group): myopic patients oldest than 10 years of age that wore single vision spectacle lenses (control group)
  Interventions: Device: Defocus Incorporated Multiple Segments (DIMS)
- Group C: patients youngest than 10 years that wear DIMS lens: myopic patients youngest than 10 years of age that wore Defocus Incorporated Multiple Segments (DIMS) spectacles
  Interventions: Device: Defocus Incorporated Multiple Segments (DIMS)
- Group D: patients youngest than 10 years (control group): myopic patients youngest than 10 years of age that wore single vision spectacle lenses (control group)
  Interventions: Device: Defocus Incorporated Multiple Segments (DIMS)

INTERVENTIONS:
Device: Defocus Incorporated Multiple Segments (DIMS) — To evaluate the effectiveness of Defocus Incorporated Multiple Segments (DIMS) in slowing myopia progression as a function of age in pediatric patients.

SUMMARY:
Purpose: To evaluate the effectiveness of Defocus Incorporated Multiple Segments (DIMS) in slowing myopia progression as a function of age in pediatric patients.

Methods: This was a non-randomized experimenter-masked retrospective controlled observational study of European individuals aged 6 -16 years with progressive myopia but no ocular pathology. The charts of the participants allocated to receive DIMS spectacles (Hoya® MiyoSmart®) or single vision spectacle lenses (control group) were retrospectively reviewed. The key outcome variables, cycloplegic spherical equivalent (SE) and axial length (AL), were measured at baseline and at 36 month follow up. The results were stratified by age into four groups: patients that wore DIMS spectacles oldest or youngest than 10 years (respectively, group A, 20 patients mean age 13.6±2.2 and group C, 20 patients mean age 9.0±1.2) and age matched control groups (group B, 18 patients mean age 13.2±2.5 and group D, mean age 8.5±0.9).

DETAILED DESCRIPTION:
Participants were allocated to the study groups, receiving DIMS spectacles, or to the control groups, wearing single vision spectacle lenses.

ELIGIBILITY:
Inclusion Criteria:

* patient age between 6-16 years
* progressive myopia with cycloplegic spherical equivalent (SE) from -0.50 to -4.00 diopters (D)
* astigmatism less than 2.50D, anisometropia under 1.25D

Exclusion Criteria:

* genetic syndromes suspected (e.g., Stickler, Marfan, etc.)
* systemic diseases
* eye diseases (such as glaucoma, juvenile cataracts, retinal abnormalities, any form of strabismus)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients with documented progressive myopiua
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
SE | 36 months
  spherical equivalent

SECONDARY OUTCOMES:
AL | 36 months
  axial lenght

CONTACTS AND LOCATIONS:
Overall Officials: Luca Buzzonetti, Principal Investigator — Bambino Gesù IRCCS Children's Hospital
Locations (1):
- Luca Buzzonetti, Rome, Italy